CLINICAL TRIAL: NCT00938327
Title: Post Marketing Surveillance to Monitor the Reactogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Oral Live Attenuated Human Rotavirus Vaccine, Rotarix™ When Administered According to the Prescribing Information to Indian Infants
Brief Title: Reactogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Rotarix™ (Human Rotavirus Vaccine) in Indian Infants
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112896
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Results first posted 2011-03-16 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2016-02

CONDITIONS: Infections, Rotavirus
Keywords: Gastroenteritis
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis | interventions — RIX4414 vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rotarix Group: Subjects who have received 2 oral doses (or a second dose for subjects who had already received the first dose prior to joining the study) of Rotarix™ at an interval of not less than 4 weeks between the doses.
  Interventions: Biological: Rotarix™

INTERVENTIONS:
Biological: Rotarix™ — Two doses of oral vaccine.

SUMMARY:
This post marketing surveillance will evaluate reactogenicity and safety data of human rotavirus vaccine when administered to healthy infants according to the Prescribing Information in India.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in this PMS.
* A male or female infant, from the age of 6 weeks at the time of the first vaccination and less than 24 weeks of age at the time of second vaccination.
* Written informed consent obtained from the parent or guardian of the subject.

Exclusion Criteria:

* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Concurrently participating in another clinical study, at any time during the surveillance period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Acute disease at the time of enrolment.
* Any history of uncorrected congenital malformation of the gastrointestinal tract that would predispose the subject for intussusception.
* Known hypersensitivity after previous administration of rotavirus vaccine or to any component of the vaccine.
* Gastroenteritis within 7 days preceding vaccination.

Ages: 6 Weeks to 167 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: subjects from the age of 6 weeks at the time of the first Rotarix™ vaccination and less than 24 weeks of age at the time of second Rotarix™ vaccination
Sampling Method: Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2009-08-03; Primary Completion 2010-02-20 (Actual); Study Completion 2010-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- India (7):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Delhi
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune

REFERENCES:
- [Background] Kumar k et al. Safety and reactogenicity of RIX4414 live attenuated human rotavirus vaccine: An Indian post-marketing surveillance study. Abstract presented at the 48th National Conference of Indian Academy of Pediatrics (Pedicon). Jaipur, India, 19-23 January 2011.
- [Background] Ruberu D et al. Post-marketing surveillance of a live-attenuated human rotavirus vaccine (Rotarix™) in India and Sri Lanka. Abstract presented at the 9th International Congress of Tropical Pediatrics (ICTP). Bangkok, Thailand, 18-20 October 2011.
- [Derived] Bravo L, Chitraka A, Liu A, Choudhury J, Kumar K, Berezo L, Cimafranca L, Chatterjee P, Garg P, Siriwardene P, Bernardo R, Mehta S, Balasubramanian S, Karkada N, Htay Han H. Reactogenicity and safety of the human rotavirus vaccine, Rotarix in The Philippines, Sri Lanka, and India: a post-marketing surveillance study. Hum Vaccin Immunother. 2014;10(8):2276-83. doi: 10.4161/hv.29280. PMID 25424932

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rotarix Group
Started | 332
Completed | 272
Not Completed | 60
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 37
Not completed — 2nd dose received outside of the study | 7
Not completed — Vaccine not received as out of stock | 9

BASELINE CHARACTERISTICS:
Arm/Group | Rotarix Group
Number analyzed (Participants) | 332
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 10.4 (4.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155
  Male | 177

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Grade 2 or 3 Symptoms (Fever, Vomiting or Diarrhoea)
Description: Grade 2 fever was defined as axillary temperature above 38.0 degrees Celsius (°C) and below or equal to 39.0°C.
  Grade 3 fever was defined as axillary temperature above 39.0°C. Grade 2 vomiting was defined as 2 episodes of vomiting per day. Grade 3 vomiting was defined as at least 3 episodes of vomiting per day. Grade 2 diarrhoea was defined as 4-5 looser than normal stools per day. Grade 3 diarrhoea was defined as at least 6 looser than normal stools per day.
Time Frame: During the 8-day (Day 0 - Day 7) follow-up period after each vaccination.
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 332
subjects | 42

2. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Cough: Cough/runny nose of any intensity Diarrhoea: Passage of three or more looser than normal stools within a day Irritability: Cried more than usual Loss of appetite: Ate less than usual Temperature: Axillary temperature greater than or equal to 37.5°C Vomiting: One or more episodes of forceful emptying of partially digested stomach contents ≥ 1 hour after feeding within a day
Time Frame: During the 8-day (Day 0 - Day 7) follow-up period after each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 332
subjects
  Cough | 43
  Diarrhoea | 14
  Irritability | 81
  Loss of appetite | 46
  Temperature (axillary) | 24
  Vomiting | 67

3. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day (Day 0 - Day 30) follow-up period after each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 332
subjects | 23

4. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Throughout the study period (from Day 0 up to Day 30)
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 332
subjects | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events: throughout the study period (Day 0-Day 30). Other adverse events: during the 8-day (Day 0-Day 7) follow-up period after each vaccination.
Arm/Group | Rotarix Group
All-Cause Mortality (participants affected / at risk) | 0/332
Serious Adverse Events (participants affected / at risk) | 0/332
Other Adverse Events (participants affected / at risk) | 133/332
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotarix Group (N=332)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 45 (55)
Decreased activity (Psychiatric disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 46 (54)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 16 (18)
Flatulence (Gastrointestinal disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Irritability (Psychiatric disorders) | 81 (97)
Lacrimation increased (Eye disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3)
Otitis media acute (Infections and infestations) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Pyrexia (General disorders) | 25 (28)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tongue discolouration (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 67 (83)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.